CLINICAL TRIAL: NCT00751504
Title: Quetiapine in the Treatment of Psychotic Depression - a Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, PD Dr. Christine Norra, MD, PhD, Prof. Dr. med. Georg Juckel, LWL University Hospital Bochum, Ruhr University of Bochum
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00040
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Psychotic Depression
Keywords: Quetiapine; Psychotic depression
MeSH Terms: interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Quetiapine — Dosage form: tablets Dosage: between 300 mg/die and 600 mg/die Frequency: once daily Duration: 6 weeks
  Other Names: Seroquel Prolong

SUMMARY:
Atypical antipsychotics have been found not only to be beneficial in the treatment of psychotic disorders, but even for depressive symptoms in patients with schizophrenia. Remarkably, preliminary data suggest that the atypical antipsychotic quetiapine has antidepressive properties. Until now, there is limited knowledge concerning the efficacy of quetiapine in major depressive illness and especially in psychotic depression. In our own clinical practice, several patients with psychotic depression were successfully treated with quetiapine as add-on therapy or as monotherapy. On the background of that, the convincing effects of quetiapine in bipolar depression, single-case reports and pilot studies concerning its effectiveness in depressive mood states in psychotic disorders as well as our clinical experiences, it is to assume that a treatment with quetiapine over a 6 weeks period show similar effects in major depressive episode with psychotic features, i.e. psychotic depression. In this pilot study we plan to investigate 20 patients with psychotic features of depression under treatment with quetiapine.

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent
* diagnosis of depression with psychotic features by DSM-IV (296.23, 296.33)
* females and males aged 18 to 65 years
* female patients of childbearing potential must be using a reliable method of contraception and have a negative pregnancy test at enrollment
* patients must be able to understand and comply with the requirements of the study
* MADRS score above 20 points

Exclusion Criteria:

* pregnancy or lactation
* any DSM-IV Axis I disorder not defined in the inclusion criteria or not in full remission
* patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* known intolerance or lack of response to quetiapine, as judged by the investigator
* use of any cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment
* use of any cytochrome P450 inducers in the 14 days preceding enrollment
* thyroid-stimulating hormone (TSH) concentration more than 10% above the upper limit of the normal range at enrollment
* administration of a depot antipsychotic injection within one dosing interval before randomisation
* substance or alcohol dependence at enrollment, as defined by DSM-IV
* opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrollment
* medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* risk of transmitting human immunodeficiency virus (HIV) or hepatitis B via blood or other body fluids
* unstable or inadequately treated medical illness, as judged by the investigator
* patients with diabetes mellitus (DM)
* an absolute neutrophil count (ANC) < 1.5x10E9 per liter
* history of idiopathic orthostatic hypotension, or condition that would predispose to
* ECG considered to show clinically significant abnormalities at enrollment as determined by a cardiologist
* involvement in the planning and conduct of the study
* previous enrollment or randomisation of treatment in the present study
* any serious and unstable somatic illness that, in the opinion of the investigator, would be negatively affects by the study medication
* participation in another drug trial within 4 weeks prior to enrollment into this study
* patients with unsufficient knowledge of the German language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
MADRS | 6 weeks

SECONDARY OUTCOMES:
Clinical laboratory evaluation | 6 weeks
Urinalysis | 6 weeks
ECG | 6 weeks
Physical and neurological examination | 6 weeks
Vital signs | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georg Juckel, M.D., Ph.D., Principal Investigator — LWL University Hospital Bochum
Locations (1):
- LWL University Hospital Bochum of the Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Adson DE, Kushner MG, Eiben KM, Schulz SC. Preliminary experience with adjunctive quetiapine in patients receiving selective serotonin reuptake inhibitors. Depress Anxiety. 2004;19(2):121-6. doi: 10.1002/da.10137. PMID 15022147
- [Background] Calabrese JR, Keck PE Jr, Macfadden W, Minkwitz M, Ketter TA, Weisler RH, Cutler AJ, McCoy R, Wilson E, Mullen J. A randomized, double-blind, placebo-controlled trial of quetiapine in the treatment of bipolar I or II depression. Am J Psychiatry. 2005 Jul;162(7):1351-60. doi: 10.1176/appi.ajp.162.7.1351. PMID 15994719
- [Background] Catapano-Friedman L. Effectiveness of quetiapine in the management of psychotic depression in an adolescent boy with bipolar disorder, mixed, with psychosis. J Child Adolesc Psychopharmacol. 2001 Summer;11(2):205-6. doi: 10.1089/104454601750284144. No abstract available. PMID 11436963
- [Background] Khouzam HR. Treatment of depressive mood in schizophrenia with the atypical antipsychotic quetiapine. Depress Anxiety. 2000;11(2):80-2. doi: 10.1002/(sici)1520-6394(2000)11:23.0.co;2-7. PMID 10812533
- [Background] Hidalgo J, Rico-Villademoros F, Calandre EP. An open-label study of quetiapine in the treatment of fibromyalgia. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jan 30;31(1):71-7. doi: 10.1016/j.pnpbp.2006.06.023. Epub 2006 Aug 4. PMID 16889882
- [Background] Masan PS. Atypical antipsychotics in the treatment of affective symptoms: a review. Ann Clin Psychiatry. 2004 Jan-Mar;16(1):3-13. doi: 10.1080/10401230490281410. PMID 15147108
- [Background] Padla D. Quetiapine resolves psychotic depression in an adolescent boy. J Child Adolesc Psychopharmacol. 2001 Summer;11(2):207-8. doi: 10.1089/104454601750284153. No abstract available. PMID 11436964
- [Background] Sajatovic M, Mullen JA, Sweitzer DE. Efficacy of quetiapine and risperidone against depressive symptoms in outpatients with psychosis. J Clin Psychiatry. 2002 Dec;63(12):1156-63. doi: 10.4088/jcp.v63n1211. PMID 12523876
- [Background] Schulz SC. New antipsychotic medications: more than old wine and new bottles. Bull Menninger Clin. 2000 Winter;64(1):60-75. PMID 10695160
- [Background] Wijkstra J, Lijmer J, Balk FJ, Geddes JR, Nolen WA. Pharmacological treatment for unipolar psychotic depression: Systematic review and meta-analysis. Br J Psychiatry. 2006 May;188:410-5. doi: 10.1192/bjp.bp.105.010470. PMID 16648526
- [Background] Zarate CA Jr, Rothschild A, Fletcher KE, Madrid A, Zapatel J. Clinical predictors of acute response with quetiapine in psychotic mood disorders. J Clin Psychiatry. 2000 Mar;61(3):185-9. doi: 10.4088/jcp.v61n0307. PMID 10817103